CLINICAL TRIAL: NCT03634904
Title: Prospective Observational Study of Serum Ceftazidime Concentrations in Hemodialysis Patients at the University Hospital of Charleroi, Belgium
Brief Title: Serum Ceftazidime Concentrations in Hemodialysis Patients
Acronym: CEFTAHEMOD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Charleroi (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Remy Demeester, Medical Doctor, Department of Internal Medicine, Centre Hospitalier Universitaire de Charleroi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUCHARLEROIPKPD001
Record Dates: First submitted 2018-08-09; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Bacterial Infections; Ceftazidime; Renal Failure Chronic Requiring Hemodialysis
Keywords: antibiotic dosing; pharmacokinetics; pharmacodynamics; hemodialysis
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug Blood sampling (Experimental): * Drug Blood sampling
  * Pharmacokinetic study measuring total and free ceftazidime concentrations
  Interventions: Drug: Drug bood sampling

INTERVENTIONS:
Drug: Drug bood sampling — Total: 6 per patient
  * after the first administration of ceftazidime (loading dose): sampling #1: at trough before 1st dialysis; sampling #2: after the end of the dialysis session;
  * after the second administration of ceftazidime (maintenance dose): sampling #3: at trough before 2d dialysis session;
  * after the third administration of ceftazidime (maintenance dose): sampling #4: at trough before 3d dialysis session;
  * after the fourth third administration of ceftazidime (maintenance dose): sampling #5: at trough before 4th dialysis session; sampling #6: after the end of the dialysis session

SUMMARY:
There is evidence that the current dosing recommendations of ceftazidime in hemodialysis patients may not reach the critical pharmacokinetic/pharmacodynamics thresholds associated with maximal efficacy.

The primary objective is to assess whether the standard doses of ceftazidime (1 or 2 g) administered at the end of the dialysis session (intermittent dialysis) allow to obtain a trough level equal or superior to 8 mg/L if the causative organism is not identified or 1 x the MIC if it is identified and its in vitro susceptibility to ceftazidime established. The secondary objectives will be (i) to assess whether a trough level equal or superior to 32 mg/L (if the causative organism is not identified) and 4 x its MIC (if identified and its in vitro susceptibility established) can be obtained; (ii) whether the criteria mentioned above also apply to the free fractions of ceftazidime; (iii) to assess whether reaching the desired free and total trough concentrations impacts the clinical outcome of the patient; (iv) to assess whether the main hemodialysis parameters impact on ceftazidime total and free serum concentrations; (v) to assess the impact of patient's residual renal function on the ceftazidime serum free and total concentrations; (vi) to assess the impact of potential drug-drug interactions on ceftazidime serum free and total concentrations; (vii) to assess how the MIC of the causative organism (if known) affects the expected effectiveness of ceftazidime.

The study will be prospective and monocentric. Drug assay will be made High Performance Liquid Chromatography (HPLC) and UV photometric detection (confirmed by tandem mass spectrometry detection[HPLC-MS-MS]). Free concentration will be measured after separation by membrane sieving.

The expected number of enrolled patients will be 20 (arbitrarily chosen but compatible with previous studies and the possibilities of the Institution in which the study will be performed. The standard dose of ceftazidime will be (i) a loading dose of 2 g followed by a maintenance dose of 1 g (the dose may be modified by the clinician in charge if deemed necessary and recorded accordingly).

The data obtained will be used for pharmacokinetic modelling and population pharmacokinetics, followed by Monte-Carlo simulations to obtain population-wide predictions and to draw conclusions that could be applicable to a larger population.

DETAILED DESCRIPTION:
Background

In case of severe infections, the first 24h of treatment are critical to limit the severity and the mortality (1). Thus, the antibiotic treatment must be initiated as soon as possible, be efficacious against the causative organism, and reach concentrations in the infected tissues larger than the minimal inhibitory concentration (MIC). In case of sepsis, pharmacokinetic parameters are modified (e.g., increase of the volume of distribution [Vd]), increase [initially] and decrease [later] of the renal clearance), which impacts on the actual concentration and activity of the antibiotic. For most antibiotics, the adaptation of the dosages is performed in a very crude fashion in case of renal failure (5). A first study has demonstrated that the antibiotic doses prescribed in case of sepsis were, in most of the cases, insufficient to obtain a concentration of 4 times or even 1 time the MIC of the causative organism during the desired fractions of the time between two successive administration (70% for ceftazidime) (6). A second study has shown that the doses of antibiotic prescribed in case of sepsis and of renal failure requiring extracorporeal hemofiltration are insufficient (7). Both studies showed also that there is a large interpatient variability in the antibiotic serum concentrations. An additional factor, rarely taken into account, is that only the free fraction of the antibiotic is active (8). Yet, the free fraction is rarely measured.

The use of ceftazidime in first intention probabilistic antibiotherapy in patients undergoing chronic hemodialysis is supported by its broad spectrum of activity against the most frequently observed organisms in this patient population, including Pseudomonas aeruginosa. The low incidence of adverse effects reported for this antibiotic makes it a better choice than ciprofloxacin. Moreover, its rather simple and controllable mode of administration (one intravenous dose administered at the end of the dialysis period) guarantees a better compliance compared to a daily oral antibiotherapy. Ceftazidime shows a low protein binding, and its activity is therefore not expected to be grossly affected in patients compared to what can be measured in vitro in reference media (9). However, mots reported data on ceftazidime protein binding have been obtained on healthy volunteers and the extent of binding of beta-lactams to serum proteins may considerably vary according to the type of subjects (10).

Presently, the recommendations for the dosages of ceftazidime in patients undergoing chronic hemodialysis are based on rather old pharmacokinetic studies assuming a plasma half-life of ceftazidime reduced to 3.3 h during hemodialysis vs. 33.6 h in anuric patients and recommending to administer half of the total daily dose at the end of the hemodialysis (11). But these recommendations do not take into account the progresses made since then in hemodialysis techniques. The international recommendations and those of the US Food and Drug Administration (FDA) recommend to administer 1 g of ceftazidime after each hemodialysis session (12). Different dialysis parameters modulating the level of removal of ceftazidime in modern dialyzers have been studied (13). This showed that the ceftazidime clearance increases with the rate of dialysis fluid flow, the ultrafiltration volume, and the urea clearance. There is a positive correlation between the increase in blood flow and the ceftazidime clearance that, however, is observed only in patients for whom an AN69 membrane was used (14). Another study has examined the impact of the use of membranes with high permeability on the pharmacodynamics of ceftazidime using mathematical modeling. This study led to a recommendation that ceftazidime should be administered at a daily dose of 1 g to obtain a serum trough concentration higher than the MIC of the causative (or suspected) organism during at least 70% of the dosing interval. A dose of 2 g of ceftazidime after each dialysis session was effective for isolates for which the MIC of ceftazidime was not superior to 16 mg/L (14). This study, however, is based on data collected in 1983 and included only 6 patients. Thus, there has been no in vivo study looking as to whether a dose of 1 or 2 g of ceftazidime administered after each dialysis session is sufficient when using contemporary dialysis equipment. Moreover, no measure of the free fraction has been made.

Objectives

The study will measure the ceftazidime serum concentrations in patients undergoing hemodialysis (before the hemodialysis session and at the end of the hemodialysis session,) and receiving standard doses of ceftazidime in order to determine whether these concentrations are sufficient based on accepted literature-based criteria concerning suspected or documented infections (15). The data will be confronted with the evolution of the patients' clinical conditions in order to draw possible correlations between these two aspects of the treatment.

Primary objective

Assess whether the standard doses of ceftazidime (1 or 2 g) administered at the end of the dialysis session (intermittent dialysis) allow to obtain the following serum concentrations:

* If the causative organism is not identified: a trough level equal or superior to 8 mg/L (1 time the MIC of the least susceptible isolates of Pseudomonas aeruginosa based on the interpretative criteria of EUCAST (European Committee on Antimicrobial Susceptibility Testing; resistance set at > 8mg/L).
* If the causative organism is identified and MIC determined and lower or equal to 8 mg/L: a trough level equal or superior to 1 time this MIC

Secondary objectives

* Assess whether the standard doses of ceftazidime (1 or 2 g) administered at the end of the dialysis session (intermittent dialysis) allow to obtain a trough concentration at 32 mg/L if the causative organism is not identified and 4 times its MIC if it is identified and its MIC determined and lower or equal to 8 mg/L
* Assess whether the criteria mentioned in the primary objectives also apply to the free fractions of ceftazidime.
* Assess whether reaching the desired free and total trough concentrations of 8 mg/L or 1 time the MIC impacts the clinical outcome of the patient (as judged by the attending physician).
* Assess whether reaching the desired free and total trough concentrations of 32 mg/L or 4 time the MIC impacts the clinical outcome of the patient (as judged by the attending physician).
* Assess the impact of main hemodialysis parameters (type of membrane, flow rate of the dialysis fluid, length of the dialysis session; volume of ultrafiltration) on the ceftazidime total and free serum concentrations.
* Assess the impact of patient's residual renal function on the ceftazidime serum free and total concentrations.
* Assess the impact of potential drug-drug interactions (based on the record of all drugs administered to the patient) impact on ceftazidime serum free and total concentrations.
* Asses how the MIC of the causative organism (if known) affects the expected effectiveness of ceftazidime, considering both the total and the free serum concentrations.

Materials and Methods

* Prospective monocentric study in the hemodialysis center of the Centre hospitalier-universitaire (CHU) of Charleroi, Belgium.
* Drug assay: all assays will be made in duplicate in two laboratories:

  * total serum concentrations in the laboratory of Biological Chemistry of the hospital where the study will be conducted (CHU) using a validated High Performance Liquid Chromatography (HPLC) separation method and an UV photometric detection
  * total and free concentrations in the laboratory of Cellular and Molecular Pharmacology of the Université catholique de Louvain (Drug Research Institute) using an HPLC separation method and a tandem mass spectrometry (MS-MS) detection method (to mitigate the risk of interferences by other drugs or metabolites in abnormal quantities). Assay of the free fraction will be made after separation by membrane sieving.
* Expected number of enrolled patients: 20. This number has been chosen arbitrarily but is compatible with (i) previous studies indicating that it is sufficient to provide useful information; (ii) the present number of patients admitted to the hospital for hemodialysis per year (from 100 to 120) with a proportion of about 20% needing antibiotic treatment for an infection for which ceftazidime is indicated.
* Sampling:

Total: 6 per patient

* after the first administration of ceftazidime (loading dose): sampling #1: at trough before 1st dialysis; sampling #2: after the end of the dialysis session
* after the second administration of ceftazidime (maintenance dose): sampling #3: at trough before 2d dialysis session
* after the third administration of ceftazidime (maintenance dose): sampling #4: at trough before 3d dialysis session
* after the fourth third administration of ceftazidime (maintenance dose): sampling #5: at trough before 4th dialysis session; sampling #6: after the end of the dialysis session

  - Ceftazidime doses
* loading dose (1st administration): 2 g
* maintenance dose (all subsequent administrations): 1 g (the dose may be modified by the clinician in charge if deemed necessary and recorded accordingly)

  * Patient's clinical and biological data collection
  * collection patient's data:
* indication(s) of ceftazidime administration
* dose and time of ceftazidime administration
* documentation of the infection and treatment outcomes: (fever (Celsius degree); suspected site (confirmed or suspected); inflammatory syndrome (biological data) (C reactive protein (mg/l), leucocytes count (/µl)); bacteriological data: clinical outcome: cure - improved - failure - relapse (by the same organism), infection-related adverse effects: septic metastasis, death; administration-related adverse effects: catheter-clogging and infection; treatment-related adverse effects: any that could be related to the drug
* parameters of the hemodialysis: type of dialysis membrane and membrane area (Polysulfone. 2 m2, 2,2m2), blood flow (ml/min (350ml/min)), dialysate flow rate (500 ml/min (fixed)), KT/V ratio (at 2d and 5th sessions) (1,2 to 1,5) where K = dialyzer clearance of urea; T= dialysis time; V = volume of distribution of urea [approximately equal to patient's total body water], access route: catheter (double lumen) or direct arterio-venous connection, length of dialysis session (minutes), added solutes (bicarbonate and other filling fluids) (mmol/liter).
* nutritional status: albumins and total proteins (g/l)
* associated medications: other antibiotics (e.g., vancomycin in case of suspicion of infection by a methicillin-resistant Gram-positive organism [e.g., S. aureus or S. epidermidis]), antivitamin K, non-steroidal anti-inflammatory agent(s).

Modeling and population pharmacokinetics Serum concentration data will be analyzed using appropriate softwares to determine the pertinent pharmacokinetic parameters for the population of patients studied. The analysis will focus on

* median and mean ceftazidime clearances and half-lives out of and during the dialysis periods
* the extraction rate of ceftazidime during the hemodialysis sessions After establishing the best model and based on Monte-Carlo simulations, the results will be used to determine whether the threshold for efficacy defined above holds true when considering the population of patients routinely undergoing hemodialysis. The general methodology and calculations approaches will be similar to those described in previous publications with adaptation if necessary (16, 17).

ELIGIBILITY:
Inclusion Criteria:

* any patient with 18 years of age or older and chronically treated by hemodialysis in the hemodialysis ward of the Institution, and
* for whom ceftazidime is administered for treating a suspected or confirmed infection for which ceftazidime is indicated, and
* who has given her/his informed consent.

Exclusion Criteria:

* patient with suspected or confirmed allergy to beta-lactam antibiotics
* pregnant women (based on patient's declaration)
* nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-15 (Estimated); Primary Completion 2020-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Trough level at 8 mg/L or 1 x the MIC | 7 days
  total trough serum concentration of ceftazidime after its administration (loading dose and maintenance dose) and determining if it is higher or equal to 8 mg/L of 1 x the MIC

SECONDARY OUTCOMES:
Trough level at 32 mg/L or 4 x the MIC | 7 days
  total trough serum concentration of ceftazidime after its administration (loading dose and maintenance dose) and determining if it is higher or equal to 32 mg/L of 4 x the MIC
Free trough level at 8 mg/L or 1 x the MIC | 7 days
  Free trough serum concentration of ceftazidime after its administration (loading dose and maintenance dose) and determining if it is higher or equal to 8 mg/L of 1 x the MIC
Free trough level at 32 mg/L or 4 x the MIC | 7 days
  Free trough serum concentration of ceftazidime after its administration (loading dose and maintenance dose) and determining if it is higher or equal to 32 mg/L of 4 x the MIC.
Impact of trough levels at 8 mg/L ot 1 x the MIC on clinical outcome | 7 days
  Number of patients for whom the total trough level is equal or higher than 8 mg/L or 1 x the MIC and who are either (i) cured, (ii) improved, or (iii) have failed to treatment (cure = cessation of the infection and no need of further treatment; improved: decrease of the signs of the infection but the same treatment is continued; failed: no cessation of the infection and need of a change of antibiotic or of its dosing).
Impact of trough levels at 32 mg/L ot 4 x the MIC on clinical outcome | 7 days
  Number of patients for whom the total trough level is equal or higher than 32 mg/L or 4 x the MIC and who are either (i) cured, (ii) improved, or (iii) have failed to treatment (cure = cessation of the infection and no need of further treatment; improved: decrease of the signs of the infection but the same treatment is continued; failed: no cessation of the infection and need of a change of antibiotic or of its dosing).
Impact of hemodialysis parameter #1 on ceftazidime total serum levels | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to the type of membrane [code no.])
Impact of hemodialysis parameter #1 on ceftazidime free serum levels | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to the type of membrane [code no.])
Impact of hemodialysis parameter #2 on ceftazidime total serum levels | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to the flow rate of the dialysis fluid [mL/min].
Impact of hemodialysis parameter #2 on ceftazidime free serum levels | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to the flow rate of the dialysis fluid [mL/min].
Impact of hemodialysis parameter #3 on ceftazidime total serum levels | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to the length of the dialysis session [min]).
Impact of hemodialysis parameter #3 on ceftazidime free serum levels | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to the length of the dialysis session [min]).
Impact of hemodialysis parameter #4 on ceftazidime total serum levels | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to the volume of ultrafiltration [L])
Impact of hemodialysis parameter #4 on ceftazidime free serum levels | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to the volume of ultrafiltration [L])
Impact of patient's residual renal function on ceftazidime total serum levels | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to their residual renal function using creatinine clearance (mL/h)
Impact of patient's residual renal function on ceftazidime free serum levels | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to their residual renal function using creatinine clearance (mL/h)
Impact of other drugs on ceftazidime serum total concentrations (mg/L). | 7 days
  Total ceftazidime concentrations (mg/L) in patients stratified according to the administration of other drugs (any)
Impact of other drugs on ceftazidime serum free concentrations (mg/L). | 7 days
  Free ceftazidime concentrations (mg/L) in patients stratified according to the administration of other drugs (any)
Impact of MIC on the clinical effectiveness of ceftazidime | 7 days
  MIC of the causative organism (if known; in mg/L) in patients stratified according to their clinical outcome (cured - improved - failed; cure = cessation of the infection and no need of further treatment; improved: decrease of the signs of the infection but the same treatment is continued; failed: no cessation of the infection and need of a change of antibiotic or of its dosing)/

CONTACTS AND LOCATIONS:
Overall Officials: Remy Demeester, MD, Principal Investigator — Centre Hospitalier Universitaire de Charleroi

REFERENCES:
- [Background] Kollef MH. Broad-spectrum antimicrobials and the treatment of serious bacterial infections: getting it right up front. Clin Infect Dis. 2008 Sep 15;47 Suppl 1:S3-13. doi: 10.1086/590061. PMID 18713047
- [Background] Wurtz R, Itokazu G, Rodvold K. Antimicrobial dosing in obese patients. Clin Infect Dis. 1997 Jul;25(1):112-8. doi: 10.1086/514505. PMID 9243045
- [Background] Falagas ME, Karageorgopoulos DE. Adjustment of dosing of antimicrobial agents for bodyweight in adults. Lancet. 2010 Jan 16;375(9710):248-51. doi: 10.1016/S0140-6736(09)60743-1. Epub 2009 Oct 28. No abstract available. PMID 19875163
- [Background] Erstad BL. Dosing of medications in morbidly obese patients in the intensive care unit setting. Intensive Care Med. 2004 Jan;30(1):18-32. doi: 10.1007/s00134-003-2059-6. Epub 2003 Nov 19. PMID 14625670
- [Background] Trotman RL, Williamson JC, Shoemaker DM, Salzer WL. Antibiotic dosing in critically ill adult patients receiving continuous renal replacement therapy. Clin Infect Dis. 2005 Oct 15;41(8):1159-66. doi: 10.1086/444500. Epub 2005 Sep 12. PMID 16163635
- [Background] Taccone FS, Laterre PF, Dugernier T, Spapen H, Delattre I, Wittebole X, De Backer D, Layeux B, Wallemacq P, Vincent JL, Jacobs F. Insufficient beta-lactam concentrations in the early phase of severe sepsis and septic shock. Crit Care. 2010;14(4):R126. doi: 10.1186/cc9091. Epub 2010 Jul 1. PMID 20594297
- [Background] Seyler L, Cotton F, Taccone FS, De Backer D, Macours P, Vincent JL, Jacobs F. Recommended beta-lactam regimens are inadequate in septic patients treated with continuous renal replacement therapy. Crit Care. 2011;15(3):R137. doi: 10.1186/cc10257. Epub 2011 Jun 6. PMID 21649882
- [Background] Zeitlinger MA, Derendorf H, Mouton JW, Cars O, Craig WA, Andes D, Theuretzbacher U. Protein binding: do we ever learn? Antimicrob Agents Chemother. 2011 Jul;55(7):3067-74. doi: 10.1128/AAC.01433-10. Epub 2011 May 2. PMID 21537013
- [Background] Lam YW, Duroux MH, Gambertoglio JG, Barriere SL, Guglielmo BJ. Effect of protein binding on serum bactericidal activities of ceftazidime and cefoperazone in healthy volunteers. Antimicrob Agents Chemother. 1988 Mar;32(3):298-302. doi: 10.1128/AAC.32.3.298. PMID 3284457
- [Background] 10. Ngougni Pokem et al. Protein binding of temocillin is lower in plasma from patients in intensive care units compared to healthy subjects: in vitro and in vivo studies ; 28th ECCMID - Session: Clinical pharmacokinetics - poster #P2219.
- [Background] Roberts JA, Ulldemolins M, Roberts MS, McWhinney B, Ungerer J, Paterson DL, Lipman J. Therapeutic drug monitoring of beta-lactams in critically ill patients: proof of concept. Int J Antimicrob Agents. 2010 Oct;36(4):332-9. doi: 10.1016/j.ijantimicag.2010.06.008. Epub 2010 Aug 3. PMID 20685085
- [Background] Nikolaidis P, Tourkantonis A. Effect of hemodialysis on ceftazidime pharmacokinetics. Clin Nephrol. 1985 Sep;24(3):142-6. PMID 3899438
- [Background] 13. GlaxoSmithKline August 2010. Fortaz (ceftazidime for injection) prescribing information. GlaxoSmithKline, Mississauga, Ontario, Canada
- [Background] Matzke GR, Frye RF, Joy MS, Palevsky PM. Determinants of ceftazidime clearance by continuous venovenous hemofiltration and continuous venovenous hemodialysis. Antimicrob Agents Chemother. 2000 Jun;44(6):1639-44. doi: 10.1128/AAC.44.6.1639-1644.2000. PMID 10817721
- [Background] Loo AS, Neely M, Anderson EJ, Ghossein C, McLaughlin MM, Scheetz MH. Pharmacodynamic target attainment for various ceftazidime dosing schemes in high-flux hemodialysis. Antimicrob Agents Chemother. 2013 Dec;57(12):5854-9. doi: 10.1128/AAC.00474-13. Epub 2013 Sep 9. PMID 24018264
- [Background] De Waele JJ, Carrette S, Carlier M, Stove V, Boelens J, Claeys G, Leroux-Roels I, Hoste E, Depuydt P, Decruyenaere J, Verstraete AG. Therapeutic drug monitoring-based dose optimisation of piperacillin and meropenem: a randomised controlled trial. Intensive Care Med. 2014 Mar;40(3):380-7. doi: 10.1007/s00134-013-3187-2. Epub 2013 Dec 20. PMID 24356862
- [Background] Vandecasteele SJ, Miranda Bastos AC, Capron A, Spinewine A, Tulkens PM, Van Bambeke F. Thrice-weekly temocillin administered after each dialysis session is appropriate for the treatment of serious Gram-negative infections in haemodialysis patients. Int J Antimicrob Agents. 2015 Dec;46(6):660-5. doi: 10.1016/j.ijantimicag.2015.09.005. Epub 2015 Oct 9. PMID 26603304
- [Background] Miranda Bastos AC, Vandecasteele SJ, Spinewine A, Tulkens PM, Van Bambeke F. Temocillin dosing in haemodialysis patients based on population pharmacokinetics of total and unbound concentrations and Monte Carlo simulations. J Antimicrob Chemother. 2018 Jun 1;73(6):1630-1638. doi: 10.1093/jac/dky078. PMID 29579214